CLINICAL TRIAL: NCT07030751
Title: Interest Of a Group-Based and Multimodal Intervention on the Quality of Life of Healthcare Students: A Randomized, Controlled, Single-Center Study.
Brief Title: Preventive Remediation for OptiMal StudentS (PROMESS-Group)
Acronym: PROMESS-Group
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROMESS-Group
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Health Behavior; Health-Related Behavior
Keywords: Health; Student; Curriculum; Behavior; Quality of life; Performance; Stress; Sleep; Fatigue; Sedentary behaviors; Physical Activity; Medical pedagogy
MeSH Terms: conditions — Health Behavior; Behavior; Fatigue; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial. Randomization into two groups: INTERVENTION group and CONTROL group (1:1). The INTERVENTION group will have the opportunity to follow a preventive remediation program based on 3 modules: stress management, sleep improvement and fatigue reduction, and sedentary behaviors reduction and physical activity promotion. The sequence of modules was established in the following order: stress module, sleep module, and physical activity module. Students in the control group will receive a specific 'compensatory' intervention after the post-intervention period.
Who Masked: Outcomes Assessor
Masking Description: Assessors of pre and posttest measures will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Interventions:
  Behavioral: Stress management, sleep improvement and fatigue reduction, sedentary behaviors reduction and physical activity promotion.
  Interventions: Behavioral: Stress management, sleep improvement and fatigue reduction, sedentary behaviors reduction and physical activity promotion.
- Control (No Intervention): Students in the control group will receive a specific 'compensatory' intervention after the post-intervention period

INTERVENTIONS:
Behavioral: Stress management, sleep improvement and fatigue reduction, sedentary behaviors reduction and physical activity promotion. — The study seeks to quantify the impact of a complex intervention based on 3 modules :
  1. Stress management
  2. Sleep improvement and fatigue reduction,
  3. Sedentary behaviors reduction and physical activity promotion.
  Students from the interventional group will follow these 3 different health-related modules in a specific order (stress, sleep, physical activity). Each module will be composed of 3 sessions. Each session includes individual interviews covering initial assessment and personalized goal setting.
  Arms: Intervention

SUMMARY:
Health students exhibit excessive sedentary behavior, elevated stress levels, and significant sleep disturbances, all of which contribute to a decline in their overall health, quality of life, and learning capacities.

The PROMESS-Group project (Preventive Remediation for OptiMal StudentS-Group) is a multimodal intervention targeting stress management, sleep improvement, and physical activity enhancement, with the aim of improving students' quality of life throughout their academic journey.

Encouraging physical activity, reducing sedentary behaviors, reducing stress, fatigue and sleep troubles during their curriculum can promote a healthier lifestyle and reduce the risk of chronic health conditions in the future.

The study seeks to quantify the impact of a complex intervention based on 3 modules (stress, sleep, physical activity) on the quality of life of health students. This study will also have a clear insight on the influence of the complex intervention on changes in stress, sleep, physical activity and sedentary behavior markers.

DETAILED DESCRIPTION:
Our project aims to help health students to adopt health-promoting behaviors during their studies in a preventive approach. This support will be provided through a multimodal intervention during their curriculum. Specifically, The PROMESS-Group program will be offered to 4th- and 5th-year medical students enrolled at the Faculties of Medicine of Lyon Est and Lyon Sud during the 2024-2025 and 2025-2026 academic years, as well as to PhD students registered in Lyon's health-related doctoral schools.

Voluntary will be randomized into 2 arms (intervention and control). Students in the control group will receive a specific 'compensatory' intervention after the post-intervention period. This intervention will be refined throughout the implementation phase and will consist of a concise yet comprehensive training covering all modules.

The intervention group will follow a preventive program based on three modules: stress management, sleep improvement and fatigue reduction, and sedentary behaviors reduction and physical activity promotion.

This program will span 16 weeks. Both groups will be characterized through a pre-post paradigm multimodal measurement. At the end of this period, we expect improvements in terms of quality of life, physical and mental health, in the interventional arm.

METHODS. POPULATION. The sample size was determined to detect a group × time interaction in a mixed linear model with random intercept for students. The variance parameters and effect size were estimated from preliminary data from a pilot study using the same model (σ²_ID = 0.315; σ²_ε = 0.162; β_interaction = 0.338), corresponding to a standardized effect of d ≈ 0.59. With a two-tailed α risk of 0.05 and 80% power, 45 students per group are required. Taking into account an expected attrition rate of 5% in the interventional group and 10% in the control group, the final size was increased to 97 students in total.

PRE-INTERVENTION. From week 1 to 2. All students will undergo a two-hour session, during which they will complete questionnaires on sedentary behavior and physical activity, stress, sleep and fatigue levels. Heart Rate Variability will be measured. Students will perform four physical fitness tests (vertical jump, maximal isometric strength, flexibility and endurance). Then, they will wear actimeters to record sleep, sedentary behaviors and physical activity levels during two weeks.

INTERVENTION. From week 3 to 14. The intervention program aims to address three key aspects of well-being. The students in the intervention group will take part in three modules, one on stress, one on sleep and fatigue, and the other on sedentary behaviors and physical activity.

The sequence of modules was established in the following order: stress module, sleep module, and physical activity module.

Each module will consist of three sessions, each lasting between 45 minutes and two hours, with approximately 10 days between each session.

To avoid too many intervention days, several sessions will be paired with another: The third stress session will be paired with the first sleep session, the second sleep session will be paired with the first physical activity session and the third sleep session will be paired with the second physical activity session.

Each session includes a period of pedagogical content delivered in small groups , as well as individual interviews between an expert and the participant (i.e.student). The sessions will be scheduled as follow:

* Session 1 Stress: Week 3
* Session 2 Stress: Week 5
* Session 3 Stress: Week 7
* Session 1 Sleep: Week 7
* Session 2 Sleep: Week 9
* Session 3 Sleep: Week 11
* Session 1 Physical activity: Week 9
* Session 2 Physical activity: Week 11
* Session 3 Physical activity: Week 13

During the interview, the expert will realize an initial assessment of student health behaviors and will give personalized goals to students. Subsequent sessions follow the same structure. Subjective and objective indicators related to each intervention domain will be recorded to assess the progress and the satsifaction of students.

POST-INTERVENTION. From week 15 to 16. All students will undergo the exact same set of measurements as described in pre-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th- or 5th-year medical student enrolled at the Faculty of Medicine (Lyon Est or Lyon Sud), or a PhD student registered in Lyon's health-related doctoral schools during the 2024-2025 or 2025-2026 academic years
* Having read the information note
* Having signed the written consent

Exclusion Criteria:

* Student who did not provide consent
* Non-French-speaking student

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Quality of life. Change from pre-intervention in a composite score obtained at the Brief Quality Of Life questionnaire at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of the quality of life is assessed four sub-scores of quality of life (i.e. physical health, psychic well-being, social relationship, environnement). The composite score is the mean of the 2 dimensions: physical health and psychological well-being.
  The measure will be done at different time frame:
  1. Pre-intervention measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  2. Post-intervention measure at week 16 : after the intervention (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score) Evolution of the 4 subscores will also be analyzed independantly.

SECONDARY OUTCOMES:
Academic self-efficacy. Change from the pre-intervention in score obtained at the General Academic Self-Efficacy Scale (GASE) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of academic self-efficacy will be assessed through the Academic self-efficacy questionnaire ranging from 5 to 20, a higher score indicating better perceived academic self-efficacy. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the intervention (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Kessler Psychological Distress Scale (KPDS). Change from the pre-intervention in score obtained at the Kessler Psychological Distress Scale (KPDS) questionnaire to the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of distress will be assessed through the Kessler Psychological Distress Scale (KPDS) questionnaire ranging from 10 (low) to 50 (extreme). The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the stress module. | Week 7
  The composite score will be the mean of two sub-scores :
  1. A stress module specific score. Mean of the scores obtained at the three 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the intervention has helped you to decrease your stress level?"
     * "Do you think the intervention allowed you to better manage the stressful events you encountered?"
  2. A stress module general score. Mean of the scores obtained at the 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?" ○ These measures will be done at the session 3 of the stress module, i.e. at week 7.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the sleep module. | Week 11
  The composite score will be the mean of two sub-scores :
  1. A sleep module specific score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the module has helped you to improve your sleep?"
     * "Do you think the module has helped you to decrease your fatigue?"
  2. A sleep module general score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?" ○ These measures will be done at session 3 of the sleep module, i.e. at week 11.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the sedentary behaviors and physical activity module. | Week 13
  The composite score will be the mean of two sub-scores :
  1. A sedentary behaviors and physical activity module specific score. Mean of the scores obtained at the three 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the module has helped you increase your level of physical fitness?")
     * "Do you think the module has helped you increase your level of physical activity?")
     * "Do you think the module has helped you decrease your level of sedentary behaviours?"
  2. A sedentary behaviors and physical activity module general score. Mean of the scores obtained at the two 100-mm VAS ranging from 0 (absolutely not) to 100 (completely) :
     * "Do you think the proposed goals were suitable for your daily life?"
     * "Do you think you can sustain the habit changes?" ○ These measures will be done at session 3 of the physical activity module, i.e. at week 13.
Perceived level of stress. Change from pre-intervention in score obtained at the Perceived Stress Scale (PSS) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of stress will be assessed through the PSS questionnaire ranging from 0 (none) to 40 (extreme). One score is assessed and can be classified as low, moderate and elevated stress. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the intervention (for the control and interventional groups).
  2. During intervention : measures will be done at week 3, 5, 7 ( for the interventional group).
  3. Post-interventional measure at week 16 : after the intervention (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Multidimensional Fatigue. Change from the pre-intervention in score obtained at the Multidimensional Fatigue Inventory (MFI) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of fatigue will be assessed through the MFI questionnaire that covers various dimensions of fatigue, including general fatigue (9 to 45), mental fatigue (6 to 30), reduced motivation (2 to 10), and reduced activity (3 to 15). The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. During intervention : measures will be done at week 7, 9, 11 (for the intervention group).
  3. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sedentary time at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. The sedentary time is the total duration of sedentary behavior, defined as periods of minimal movement or activity, measured in minutes/day.
  The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.0 ○ Change = (Week 16 score - Week 1 score)
Coping strategies. Change from pre-intervention in scores obtained at the Brief Cope Inventory (BCI) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students' coping strategies (social support, active resolution, positive thinking, and avoidance) will be assessed through the BCI questionnaire, each score ranging from 1 to 4; a high score indicating the behaviour was highly engaged. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. During intervention : measures will be done at week 3, 5, 7 (for the interventional group).
  3. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Perceived level of sleep troubles. Change from pre-intervention in score obtained at the Pittsburgh Sleep Questionnaire Inventory (PSQI) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of sleep troubles will be assessed through the PSQI score ranging from 0 (none) to 21 (extreme). This score classified the presence or absence of sleep troubles. It can be divided into eight sub-scores (i.e., sleep quality, sleep latency, time spent in bed, sleep time, habitual sleep efficiency, sleep disturbance, use of sleeping medication and daytime dysfunction).
  The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. During intervention : measures will be done at week 7, 9, 11 (for the interventional group).
  3. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Moderate-to-vigorous Physical Activity (MVPA) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. MVPA refers to physical activities that require moderate to high levels of effort and significantly increase heart rate and breathing. These activities contribute to improved cardiovascular health, fitness, and overall well-being. MVPA encompasses a range of activities that are more intense than sedentary behaviors but less intense than vigorous activities. MVPA is measured in minutes/day. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control a
Heart rate variability (HRV) marker. Change from pre-intervention in the RMSSD score in at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physiological stress will be assessed through the RMSSD, an HRV marker. RMSSD is the most commonly measured form of HRV, it calculates the difference between successive inter-beat-intervals (IBI) in ms, squares these values and takes the root of the mean. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
  3. The measure will be done every 2 weeks from February to July in the intervention group, i.e. at week 1, 3, 5, 7, 9, 11, 13, 16 ○ Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep regularity index at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep regularity index is a measure that evaluates the consistency of an individual's sleep habits over a given period. It takes into account the regularity of bedtime and wake-up times on a daily basis. The higher the sleep regularity index, the more consistent and regular the individual's sleep habits are considered to be. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in VO2max through the endurance test at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). During this test, the velocity at maximal aerobic (VMA) is the maximum speed (velocity) reached where the individual can still maintain aerobic metabolism without transitioning into anaerobic metabolism. VO2max refers to the maximum rate of oxygen consumption during intense exercise, typically measured in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). It is a key indicator of an individual's cardiovascular fitness and aerobic endurance. The VO2max was estimated as 3.5 times VMA. The VO2max through the endurance will be recorded at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
VAS - stressors quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived quantity of stressors. | Week 3, 5, 7
  The students quantity of stressors will be assessed on a 100-mm Visual Analogue Scale (VAS: "In the past two weeks, how many stressful situations have you encountered?") ranging from 0 (maximum/extreme) to 100 (zero). The measure will be done in the intervention group, i.e. at week 3, 5, 7.
VAS - stress quality: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the emotional valence associated with the stress level. | Week 3, 5, 7
  The emotional valence associated of the students stress level will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your stress?") ranging from 0 (very negative feelings) to 100 (very positive feelings). The measure will be done in the intervention group, i.e. at week 3, 5, 7.
VAS - stress coping. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the management of stressful situations. | Week 3, 5, 7
  The students management of stressful situations will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how did you manage your stressful situations?") ranging from 0 (very bad stress coping) to 100 (excellent stress coping). The measure will be done in the intervention group, i.e. at week 3, 5, 7.
VAS - stress quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of stress. | Week 3, 5, 7
  The student's level of stress will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your stress level?") ranging from 0 (total absence of stress) to 100 (stress maximal). The measure will be done in the intervention group, i.e. at week 3, 5, 7.
VAS - sleep quality. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) characterizing the sleep quality. | Week 7, 9, 11
  The students' level of sleep quality will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (the worst quality of sleep possible) to 100 (the best quality of sleep possible). The measure will be done in the intervention group, i.e. at week 7, 9, 11.
VAS - sleep quantity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the quantity of sleep. | Week 7, 9, 11
  The student level of sleep quantity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (quantity of sleep largely insufficient) to 100 (quantity of sleep largely sufficient). The measure will be done in the intervention group, i.e. at week 7, 9, 11.
VAS - sleep fatigue. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of fatigue. | Week 7, 9, 11
  The student's level of fatigue will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your physical and mental fatigue levels ?") ranging from 0 (extreme fatigue) to 100 (absence total of fatigue). The measure will be done in the intervention group, i.e. at week 7, 9, 11.
VAS - physical fitness. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of physical fitness. | Week 9, 11, 13
  The students' level of physical fitness will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical fitness?") ranging from 0 (bad shape) to 100 (best shape ever). The measure will be done every 2 weeks in the intervention group, i.e. at week 9, 11, 13.
VAS - physical activity. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the level of physical activity. | Week 9, 11, 13
  The student's level of physical activity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of physical activity?") ranging from 0 (completely inactive) to 100 (extremely active). The measure will be done every 2 weeks in the intervention group, i.e. at week 9, 11, 13.
VAS - sedentary behaviors. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of sedentary behaviors. | Week 9, 11, 13
  The students level of sedentary behaviors will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your level of sedentary behaviors?") ranging from 0 (extremely sedentary) to 100 (absolutely not sedentary). The measure will be done every 2 weeks in the intervention group, i.e. at week 9, 11, 13.
Epworth Sleepiness scale. Change from the pre-intervention in score obtained at the Epworth Sleepiness scale at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of diurnal sleepiness will be assessed through the Epworth Sleepiness scale ranging from 0 (none) to 24 (extreme). The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Perceived level of physical activity. Change from the pre-intervention in score obtained at the Rapid Assessment of Physical Activity (RAPA) questionnaire to the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student level of physical activity will be assessed through the RAPA questionnaire. Level of physical activity, including aerobic, strength, and flexibility is self-assessed. Scores are expressed in hours per day for week and weekend days. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. During the intervention : measures will be done at week 9, 11, 13 (for the interventional group).
  3. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Perceived level of physical activity and sedentary. Change from the pre-intervention in score obtained at the Onaps-PAQ questionnaire to the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of physical activity and sedentary will be assessed through the Onaps-PAQ (National Observatory for Physical Activity and Sedentariness - Physical Activity Questionnaires) during a typical week. Scores are expressed in hours per day for week and weekend days. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. During the intervention : measures will be done at week 9, 11, 13 (for the interventional group).
  3. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Loneliness scale (ESUL). Change from the pre-intervention in score obtained at the Loneliness scale (ESUL) to the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of loneliness will be assessed through the Loneliness scale (ESUL) questionnaire ranging from 20 (low) to 80 (extreme). The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
ASSIST-Lite (Alcohol, Smoking and Substance Involvement Screening Tool - Lite). Change from the pre-intervention in score obtained at the ASSIST-Lite (Alcohol, Smoking and Substance Involvement Screening Tool-Lite) questionnaire to the post-intervention | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of substances use will be assessed through the ASSIST-Lite (Alcohol, Smoking and Substance Involvement Screening Tool - Lite). questionnaire ranging from 20 (low) 80 (extreme). The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in cardiac coherence at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physiological stress will be assessed through cardiac coherence, an HRV marker. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
  3. The measure will be done every 2 weeks from February to July in the intervention group, i.e. at week 1, 3, 5, 7, 9, 11, 13, 16 ○ Change = (Week 16 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in the SDNN score at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physiological stress will be assessed through the SDNN score, an HRV marker. SDNN is the standard deviation of the inter-beat-intervals (IBI) measured in ms, NN means "normal" beats, i.e, removing abnormal or false beats.The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
  3. The measure will be done every 2 weeks from February to July in the intervention group, i.e. at week 1, 3, 5, 7, 9, 11, 13, 16 ○ Change = (Week 16 score - Week 1 score)
Heart rate variability (HRV) marker. Change from pre-intervention in the pnn50% score in at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physiological stress will be assessed through the pnn50%, an HRV marker. NN50 is the Number of pairs of successive intervals that differ by greater than 50ms. And pNN50 which is more typically used is the proportion of NN50 over all N-N intervals in a sample, expressed as a percentage.The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
  3. The measure will be done every 2 weeks from February to July in the intervention group, i.e. at week 1, 3, 5, 7, 9, 11, 13, 16 ○ Change = (Week 16 score - Week 1 score)
Heart rate variability (HRV) markers.Change from pre-intervention in the Low frequency / High frequency ratio (LF/HF) ratio in at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The students level of physiological stress will be assessed through the LF/HF ratio, an HRV marker. The HF band is typically correlated with RMSSD and NN50, lower HF power is associated with stress and anxiety. It is primarily associated with activity in the parasympathetic nervous system. The LF band is typically associated with the sympathetic nervous system and the HF/LF ratio is often used as a measure of sympathetic-parasympathetic balance in the nervous system. The measures will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
  3. The measure will be done every 2 weeks from February to July in the intervention group, i.e. at week 1, 3, 5, 7, 9, 11, 13, 16 ○ Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Time in Bed at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings.The time in bed (in hours/day) refers to the total duration between the time an individual gets into bed with the intention of sleeping and the time he/she get out of bed. It includes both the time spent asleep (total sleep time) and any periods of wakefulness while in bed. Essentially, it represents the total time allocated for sleep, regardless of whether the individual is actually sleeping during that time. The measure will be done at different time frames:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups) for a measuring period of 2 weeks.
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Total Sleep duration at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students level of sleep will be accessed through the actimetry recordings. The total duration of sleep is obtained during a specified period, measured in hours/day. It represents the overall quantity of sleep obtained by an individual.The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep efficiency at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' level of sleep will be accessed through the actimetry recordings.The sleep efficiency is the ratio of total sleep time to the total time spent in bed, expressed as a percentage. It reflects how effectively one is sleeping during the time allotted for sleep. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Onset Latency at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' level of sleep will be accessed through the actimetry recordings. The sleep onset latency is the amount of time it takes for an individual to fall asleep after getting into bed, measured from the time the lights are turned off until sleep onset, reported in minutes.The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Wake after Sleep Onset at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' level of sleep will be accessed through the actimetry recordings.The wake after sleep onset measures the total amount of time spent awake after initially falling asleep, reported in minutes. It reflects the disruptions in sleep continuity. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Number of Awakenings at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' level of sleep will be accessed through the actimetry recordings.The number of awakenings represents the frequency of brief awakenings during the sleep period. Each awakening may disrupt the continuity of sleep and impact sleep quality. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Mid-sleep point at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' level of sleep will be accessed through the actimetry recordings.The mid-sleep point refers to the midpoint of an individual's sleep period. It is calculated by finding the halfway point between the time of sleep onset (when the individual falls asleep) and the time of sleep offset (when the individual wakes up). The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Bedtime at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' basal level of sleep will be accessed through the actimetry recordings. The bedtime is the time at which an individual goes to bed with the intention of sleeping.The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Onset time at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep onset time refers to the time at which an individual falls asleep after initially getting into bed with the intention of sleeping, measured in minutes. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Sleep Inertia at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' basal level of sleep will be accessed through the actimetry recordings. The sleep inertia refers to the periods between wake-up time and get-up time, measured in minutes. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in Wake-up time at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' basal level of sleep will be accessed through the actimetry recordings. The wake-up time refers to the time at which an individual awakens from sleep in the morning. The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in light physical activity at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Light physical activity refers to any activity that requires minimal effort and only slightly elevated heart rate and breathing, measured in minutes/day. It involves movement that is more than sedentary behavior but does not reach the intensity level of moderate-to-vigorous physical activity (MVPA). Light physical activities are typically those that can be performed during daily tasks or leisurely pursuits and do not typically lead to significant sweating or increased breathing rate.The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post
Actimetry records. Change from pre-intervention in sedentary breaks at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Sedentary breaks refer to short periods of time during which individuals interrupt prolonged sitting or sedentary behavior by engaging in light physical activity or standing.
  The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Actimetry records. Change from pre-intervention in prolonged sedentary bouts at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The objective students' levels of physical activity and sedentary behavior will be accessed through the actimetry recordings. Prolonged sedentary bouts refer to extended periods of time during which individuals engage in minimal physical activity or remain in a seated or reclined position without interruption. These bouts typically last for prolonged durations, measured in minutes/day, often exceeding 30 minutes or more at a time.The measure will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups) for a measuring period of 2 weeks.
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Strength. Change from pre-intervention in the force developed during a maximal isometric contraction of the quadriceps at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a muscular strength test.
  The maximum isometric strength of the quadriceps during the strength test will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in height of jump at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The squat jump is plyometric exercise in which a person bends their knees to lower their body into a squat position, then performs an explosive jump upwards by extending the hips, knees, and ankles simultaneously. During this exercise, the height of jump will be measured (in cm).
  The high of jump will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in time of flight at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the time of flight will be measured (in seconds).
  The time of flight will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Power. Change from pre-intervention in relative power at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a power test, a vertical jump. During this exercise, the relative power can be estimated. The relative power will be done at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in speed through the endurance test at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The speed through the endurance will be recorded at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Endurance. Change from pre-intervention in heart rate during the endurance test at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The heart rate will be measured at three moments: maximum, submaximal, at 1 minute, and 3 minutes of recovery. The measure will be recorded at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Flexibility. Change from pre-intervention in flexibility at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of flexibility will be assessed through the Sit and Reach Test. During this exercise, the flexibility of the lower back and hamstrings can be measured. The flexibility of the lower back and hamstrings will be done (in cm) at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Physical fitness markers - Flexibility. Change from pre-intervention in flexibility at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The student's level of flexibility will be assessed through the Shoulder Flexibility Test. During this exercise, the flexibility of the shoulders can be measured. The flexibility of the shoulders will be done (in cm) at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Body composition markers. Change from the pre-intervention in Body Mass Index (BMI) at the post-interventional measure at Week 16. | Week 1 (Pre-intervention) and Week 16 (Post-intervention)
  The BMI is a measure used to assess an individual's body weight in relation to their height. It's calculated by dividing a person's weight in kilograms by the square of their height in meters (BMI = weight in kilograms / (height in meters)²). BMI provides a general indication of whether a person's weight falls within a healthy range relative to their height. Here's how BMI categories are typically interpreted:
  Underweight: BMI less than 18.5 Normal weight: BMI between 18.5 and 24.9 Overweight: BMI between 25 and 29.9 Obesity: BMI 30 or greater
  The measure will be recorded at different time frame:
  1. Pre-interventional measure at week 1: before any involvement in the modules (for the control and interventional groups).
  2. Post-interventional measure at week 16 : after the modules (for the control and interventional groups).
     * Change = (Week 16 score - Week 1 score)
Question recommendation. Answer to the question "Would you recommend a friend to participate in the PROMESS-group project?" asked during the post-intervention. | Week 16 (Post-intervention)
  "Would you recommend a friend to participate in PROMESS-group?" The answer may be YES or NO. This will provide information on students' willingness to recommend the project and may represent their overall perception and appreciation of the project. This measure will be done during the post-interventional period at week 16 (for the control and interventional groups).
Question change of habits. Answer to the question "Do you think that your participation in the PROMESS-group project has modified your health behaviors/actions?" asked during the post-intervention. | Week 16 (Post-intervention)
  "Health behavior refers to all individual actions and habits that have an impact on health, including lifestyle choices, hygiene practices, diets, physical activity, sleep, use of substances such as tobacco and alcohol, stress management and compliance with medical recommendations. These behaviors play a crucial role in disease prevention, health promotion and overall well-being. Based on this definition, do you think that your participation in the PROMESS-group project has modified your health behaviors/actions?". The answer can be YES or NO.This measure will be done during the post-interventional period at week 16 (for the control and interventional groups).
Question change of habits. Answer to the question ""For which behaviors do you think you have modified your habits/actions?" asked during the post-intervention. | Week 16 (Post-intervention)
  If the student answers yes at the previous question ("Do you think that your participation in the PROMESS-group project has modified your health behaviors/actions?"), he/she will be asked: "For which behaviors do you think you have modified your habits/actions?". They may answer YES (positive changes), YES (negative change), NO (no change for this behavior) among a pre-established list of behaviors (stress, sleep, sedentary or physical activity behaviors). They may also declare additional different habits changes. This measure will be done during the post-interventional period at week 16 (for the control and interventional groups).
Quantity of stressors. Score obtained at the Holmes and Rahe Questionnaire Inventory during the pre-intervention. | Week 1 (Pre-intervention)
  The quantity of stressors met by students during the last years will be assessed with the Holmes and Rahe Questionnaire inventory. One score is assessed and can be classified as low, medium and high risk of health degradation. This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).
Big-5. Scores obtained at the Big-5 questionnaire. | Week 1 (Pre-intervention)
  The students personality traits (i.e. agreeableness, openness, consciousness, extraversion, neuroticism) will be assessed through the Big-5 questionnaire. Each score ranges from one to five. This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).
Composite Scale of Morningness. Score obtained at the Composite Scale of Morningness (CSM). | Week 1 (Pre-intervention)
  The students chronotype are assessed through the CSM. A total score can also be assessed (from 13 to 55). A score of 22 or less indicates an evening chronotype, a score above 44 indicates a morning chronotype, and scores in between receive an intermediate classification. This measure will be done during the pre-interventional period at week 1 (for the control and interventional groups).

CONTACTS AND LOCATIONS:
Locations (1):
- Research on Healthcare Performance Lab U1290, Lyon, France

IPD SHARING:
Plan to Share IPD: No